CLINICAL TRIAL: NCT03951792
Title: Time Longitudinal Study of the Microbiome in Colorectal Cancer Subjects
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 21-001536; R01CA179243 (NIH); 18-009965 (Other: Mayo Clinic in Rohester); P30CA015083 (NIH)
Record Dates: First submitted 2019-05-14; First posted 2019-05-15 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Cancer Colon; Gastrointestinal Disease
MeSH Terms: conditions — Colonic Neoplasms; Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue Biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colorectal Cancer Subjects: Subjects under going colorectal resection with colorectal cancer will have tissue and stool collected
- Benign Colon Resection Subjects: Subjects under going colorectal resection without colorectal cancer will have tissue and stool collected

SUMMARY:
Researchers are trying to determine whether certain microbiome cause cancer or whether they are part of the microbiome in the gut due to the presence of cancer.

DETAILED DESCRIPTION:
The purpose of this research is to learn about how the gastrointestinal bacteria (microbiome) can contribute to colon cancer, and how it may change due to colon cancer. In addition, we are going to study the features of the microbiome that can help predict recovery after colon resection. To do this, we are going to compare the microbiome from subjects with colon cancer to subjects without colon cancer.

Study participation involves collection of stool samples before and after your surgery, as well as samples of residual (left-over) colon tissue from your surgery. We would also like to collect optional samples from your follow-up colonoscopy. You may be in the study for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients undergoing bowel resection by any standard surgical approach.

Exclusion Criteria:

* Female that are pregnant
* Currently receiving or have received pelvic cancer radiation therapy in the past 2 weeks.
* Currently receiving or have received chemotherapy in the past 2 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing bowel resection by any standard surgical approach at Mayo Clinic in Rochester, MN.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
DNA/RNA Biomarkers | 5 years
  Biomarkers will be defined by extracting DNA/RNA from tissue biopsies and stored for specific gene extractions.
Microbial 16S rDNA Biomarkers | 5 years
  The samples will be used to partially (V3-V5 region) amplify the microbial 16S rDNA genes through a polymerase chain reaction (PCR). The PCR product will subsequently be purified and quantified before being sequenced. They will also be used for whole genome sequencing (WGS) and Methylation sequencing (Methyl-Seq). The RNA will be used for RNAseq.

SECONDARY OUTCOMES:
Protein Measurements | 5 years
  Based on our initial findings protein measurements may also be performed on any extra residual specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas L. Chia, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials